CLINICAL TRIAL: NCT00271518
Title: A Phase III, Multi-centre, Randomised, Parallel Group Study of Safety and Efficacy of the LB03002 a New Sustained Release Formulation of Human Recombinant Growth Hormone as Compared to Standard Daily Therapy in Treatment Naive Children With Growth Failure Due to Insufficient Secretion of Endogenous Growth Hormone
Brief Title: Treatment of Children With Insufficient Secretion of Growth Hormone
Acronym: BPLG-004
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: LG Life Sciences (Industry)
Collaborators: BioPartners GmbH (Industry)
Responsible Party: Songmi Lee/Clinical Research Manager, LG Life Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPLG-004
Expanded Access: Available
Record Dates: First submitted 2005-12-29; First posted 2006-01-02 (Estimated); Last update posted 2010-03-17 (Estimated); Status verified 2010-03

CONDITIONS: Growth Hormone Deficiency (GHD)
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — Growth Hormone; Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LB03002, sustained release human hGH (Experimental): LB03002
  Interventions: Drug: growth hormone (somatropin)

INTERVENTIONS:
Drug: growth hormone (somatropin) — dosing regimen is weight based.

SUMMARY:
The purpose of this study is to compare a new weekly administered growth hormone preparation with standard daily treatment in children with insufficient secretion of growth hormone

DETAILED DESCRIPTION:
Treatment with recombinant human growth hormone (somatropin) has been proven to be effective in stimulating height velocity and improving height in children with short stature due to insufficient endogenous Growth Hormone secretion. Currently somatropin is available in daily injection formulations. The requirement of daily administration causes significant burden and interruption of normal daily life. A product with less frequent dosing regimen will provide considerable improvement over currently available conventional replacement therapy regimens.

The primary objective of this study is to demonstrate the clinical comparability in terms of safety and efficacy of a new sustained release recombinant human growth hormone formulation to that of daily growth hormone.

ELIGIBILITY:
Inclusion Criteria:

* Pre-pubertal children (boys age: > 3 and <12 years or girls: age >3 and <11 years) with isolated GH insufficiency, GH insufficiency as part of multiple pituitary hormone deficiencies, or organic GH insufficiency. If GH insufficiency occurred after treatment for any brain tumour, the patient has to be at least one year in clinical remission which has to be confirmed by computer tomography (CT) or magnetic resonance imaging (MRI) scan (with contrast) within 3 months prior to study entry
* Children with negative signs for intracranial tumour or tumour growth as confirmed with a CT or MRI scan (with contrast) within 12 months prior to inclusion or at inclusion visit
* Confirmed diagnosis of GH insufficiency as determined by two different GH provocation tests, defined as a peak plasma GH level of ≤7 ng/ml
* No prior exposure to rhGH therapy (GH-treatment naive)
* Height (HT), except in children suffering from organic GH insufficiency, of at least 2.0 standard deviations (SD) (HT SDS £-2.0) below the mean height for chronological age (CA) and sex according to the 2000 standards from the Centers for Disease Control and Prevention (CDC).
* Height velocity (HV) of at least 1 SD (HV SDS £-1) below the mean HV for CA and sex according to the standards of Prader. The minimum time between two standard height measurements should be at least 6 month before inclusion.
* Baseline IGF-I level of at least 0.5 SD (IGF-1 SDS£-0.5) below the mean IGF-1 level standardised for age and sex according to the central laboratory reference values.
* Written informed consent of parent or legal guardian of subject.

Exclusion Criteria:

* Any clinically significant abnormality likely to affect growth or the ability to evaluate growth, such as, but not limited to, chronic diseases like renal insufficiency, spinal cord irradiation, and malnutrition (BMI must be above -2SD and below +2SD of mean BMI for the chronological age and sex according to the CDC standards, and albumin must be above lower limit of normal (LLN) of the central laboratory for a patient to be included).
* Patients with overt diabetes mellitus (Fasting blood sugar >126 mg/dl) and impaired fasting sugar (Fasting blood sugar >100 mg/dl after repeated blood analysis)
* Chromosomal abnormalities and medical "syndromes" (Turner's syndrome, Laron syndrome, Noonan syndrome or absence of growth hormone receptors), with the exception of septo-optic dysplasia
* Congenital abnormalities (causing skeletal abnormalities), Russell-Silver Syndrome, skeletal dysplasias
* Closed epiphyses
* Other growth promoting medication such as anabolic steroids, with the exception of pituitary hormone replacement therapy, thyroxine, hydrocortisone and desmopressin (DDAVP) replacement therapies
* Children requiring glucocorticoid therapy (e.g. asthma) that are on the dose of more than 400 µg/d of inhaled budesonide or equivalents inhaled for longer than 1 month during a calendar year
* Bone age (BA) higher than chronological age
* Poorly controlled or uncontrolled pituitary insufficiencies of other axes (e.g., thyroid-stimulating hormone, adrenocorticotropic hormone/cortisol, vasopressin deficiency): Children who are on stable replacement therapy for less than 6 months for thyroid replacement therapy, and less than 3 months for other hormonal deficiencies prior to enrolment
* Major medical conditions and/or presence of contraindication to rhGH treatment
* Known or suspected HIV-positive patient or patient with advanced diseases such as AIDS or tuberculosis
* Drug, substance, or alcohol abuse
* Known hypersensitivity to the components of study medication
* Evidence of tumour growth or malignant disease
* Presence of anti-hGH antibodies at screening
* The patient and/or the parent/legal guardian are likely to be non-compliant in respect to study conduct.

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 144 (Estimated)
Dates: Start 2005-09; Primary Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Height velocity at the end of 12 months treatment | 12 months

SECONDARY OUTCOMES:
1.Height velocity SD score (HV SDS) after 12 months treatment, 2.Serum IGF-I levels3. Serum IGFBP-3 levels | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology, Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Khadilkar V, Radjuk KA, Bolshova E, Khadgawat R, El Kholy M, Desai M, Peterkova V, Mericq V, Kratzsch J, Siepl EC, Martin D, Lopez P, Ji HJ, Bae YJ, Lee JH, Saenger PH. 24-month use of once-weekly GH, LB03002, in prepubertal children with GH deficiency. J Clin Endocrinol Metab. 2014 Jan;99(1):126-32. doi: 10.1210/jc.2013-2502. Epub 2013 Dec 20. PMID 24170106